CLINICAL TRIAL: NCT05454839
Title: Preferences for Services in a Patient's First Six Months on Antiretroviral Therapy for HIV in South Africa
Acronym: PREFER-SA
Status: Active, not recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: University of the Witwatersrand, South Africa (Unknown); Clinton Health Access Initiative Inc. (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: H-42726
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: HIV; antiretroviral treatment; differentiated service delivery; retention in care
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Adult patients within 6 months of ART initiation or re-initiation
  Interventions: Other: Survey; Other: Focus group

INTERVENTIONS:
Other: Survey — Interviewer-administered survey
Other: Focus group — Focus group for selected participants

SUMMARY:
With the advent of universal eligibility for HIV treatment ("treat all") and same-day and community-based antiretroviral therapy (ART) initiation, retention in care after a patient has started ART remains the main challenge to achieving optimal outcomes in HIV treatment programs. Consistently across both time and geography, the highest risk for loss from care is during a patient's first six months after ART initiation, with about quarter of all patients not retained by the end of month 6.

One of the reasons for the high attrition from care in this early retention period is that the model of care offered to most newly-initiating and re-initiating patients has barely evolved from its original outlines. Patients in their first six months on ART are generally not eligible for lower-intensity, patient-centered "differentiated service delivery" models that make remaining in care easier for experienced patients. Instead, most early patients must still make multiple clinic visits that include clinical consultations with providers, and most can receive only 1-2 month supplies of medications at a time.

This protocol is for the PREFER-South Africa study, an activity of the Retain6 project. Retain6 aims to develop new models of care for patients' first six months on ART. PREFER-South Africa will collect data on patients' characteristics, clinical and non-clinical needs, and preferences for different types of services during their first six months after initiating ART. The investigators will conduct an observational, prospective cohort survey of newly-initiated or re-initiated adult ART patients at a selected set of 18 healthcare facilities in South Africa. Results are expected to inform the design of better models of service delivery for the early treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV and on ART for 0-6 six months at the study site
* ≥ 18 years old (18 and older considered adult for research purposes in South Africa)
* Presented at the study site for routine HIV-related care
* Provide written informed consent to participate.
* For patients providing a dried blood spot specimen, initiating or re-initiating ART at the study enrollment visit.

Exclusion Criteria:

* Unable to communicate in any of the languages into which the questionnaire has been translated or that is known to the research assistant
* Not physically, mentally, or emotionally able to participate in the study, in the opinion of the investigators or study staff
* Unwilling to take the time required to complete the questionnaire on the day of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have initiated or re-initiated antiretroviral therapy for HIV within 6 months of study enrollment, including the same day.
Sampling Method: Non-Probability Sample
Enrollment: 1098 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Retention | 6 months
  Not missing a scheduled clinical or medication pickup visit during the first 6 months after treatment initiation by more than 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Rosen, Study Director — Boston University
Locations (2):
- Mhairi Maskew, Johannesburg, Gauteng, South Africa
- Clinton Health Access Initiative, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided
Will share anonymized data that are generated by the study. Medical record data will not belong to the study team.

REFERENCES:
- [Background] Rosen S, Grimsrud A, Ehrenkranz P, Katz I. Models of service delivery for optimizing a patient's first six months on antiretroviral therapy for HIV: an applied research agenda. Gates Open Res. 2020 Jul 29;4:116. doi: 10.12688/gatesopenres.13159.1. eCollection 2020. PMID 32875281
- [Background] Maskew M, Ntjikelane V, Juntunen A, Scott N, Benade M, Sande L, Hasweeka P, Haimbe P, Lumano-Mulenga P, Shakewelele H, Mukumbwa-Mwenechanya M, Rosen S. Preferences for services in a patient's first six months on antiretroviral therapy for HIV in South Africa and Zambia (PREFER): research protocol for a prospective observational cohort study. Gates Open Res. 2024 Jan 9;7:119. doi: 10.12688/gatesopenres.14682.2. eCollection 2023. PMID 38343769
- [Derived] Benade M, Maskew M, Ntjikelane V, Scott N, Ngcobo N, Nichols B, Malala L, Manganye M, Rosen S. Prior antiretroviral therapy exposure among clients presenting for HIV treatment initiation in South Africa: an exploratory mixed-methods study using multiple indicators of exposure. BMC Infect Dis. 2025 Jul 26;25(1):947. doi: 10.1186/s12879-025-11340-4. PMID 40713520
- [Derived] Mutanda N, Morgan A, Kamanga A, Sande L, Ntjikelane V, Maskew M, Haimbe P, Lumano-Mulenga P, Rosen S, Scott N. Experiences and Preferences in Zambia and South Africa for Delivery of HIV Treatment During a Client's First Six Months: Results of the PREFER Study's Cross-Sectional Baseline Survey. AIDS Behav. 2025 Jun;29(6):1713-1728. doi: 10.1007/s10461-025-04640-y. Epub 2025 Feb 1. PMID 39891834